CLINICAL TRIAL: NCT00036036
Title: Phase II Study of CP-461 in Patients With Advanced Renal Cell Cancer
Brief Title: Study of CP-461 in Patients With Advanced Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-461-003
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Renal Cell Carcinoma
Keywords: renal; renal cell cancer; renal cell carcinoma; kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — (5-fluoro-2-methyl-1-(4-pyridyl)methylene-3-(N-benzyl)-indene)-acetamide hydrochloride

INTERVENTIONS:
Drug: CP-461

SUMMARY:
The purpose of this study is to determine the efficacy of CP-461 given twice-daily orally in locally advanced or metastatic renal cell cancer and to evaluate the safety profile of CP-461 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Measurable metastatic or locally advanced disease.
2. Histologically confirmed renal cell cancer.
3. No radiotherapy within 4 weeks prior to entering the study. No more than 1 prior systemic therapy for advanced disease. Prior adjuvant systemic therapy is allowed. Patients must have fully recovered from the acute effects of prior therapy.
4. Expected remaining life span > or = three months.
5. ECOG performance status 0-2.
6. > or = 18 years of legal age.
7. Male patients, or non-pregnant and non-lactating female patients who are either using adequate birth control, surgically sterile or post-menopausal.
8. Negative serum pregnancy test, if fertile female.
9. Willingness and ability to sign an informed consent document.

Exclusion Criteria:

1. Uncontrolled or symptomatic brain metastases.
2. Use of an investigational medication or device within one month of initiating study therapy.
3. Absolute granulocyte count < or = 1500/mm3; Platelet count < or = 100,000/mm3; total serum bilirubin above the upper limit of normal; serum creatinine > or = 2.2 mg/dL; AST/ALT > 2.5 ULN.
4. Any condition or any medication which may interfere with the conduct of the study.
5. Current active malignancy other than renal cell cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2001-07; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States